CLINICAL TRIAL: NCT01540006
Title: Outpatient Cardiac Rehabilitation in Austria
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Head of institute, Paracelsus Medical University
Other Study IDs: UISM-6
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Physical activity — 50min of endurance training combined with 45min of calisthenics; 1-3x/week; 6-24 weeks

SUMMARY:
The aim of this prospective trial is the manifestation of guidelines developed for outpatient cardiac rehabilitation in Austria.

The evaluation of prospective and retrospective data is supposed to give evidence on morbidity and/or mortality advantages compared to patients not participating in cardiac rehabilitation programs.

The database created in this context is supposed to pave the way as instrument to document and comprehend quality and cost effectiveness of outpatient cardiac rehabilitation in Austria as a key for quality management.

ELIGIBILITY:
Inclusion Criteria:

* heart disease

Exclusion Criteria:

* participation in another study within the previous 6 months
* Medical conditions which prevent patients from complying with the exercise program
* Acute infections
* Hypertrophic cardiomyopathy
* Pulmonary artery embolism or phlebothrombosis within the previous 6 months
* Unstable angina pectoris
* Heart failure (NYHA IV)
* Hemodynamically unstable arrhythmia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients with heart disease willing to participate in an ambulant cardiac rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Physical work capacity (PWC) | 6 weeks
  PWC is measuered by gradded exercise test on cycling ergometer before and after rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Josef Niebauer, MD, PhD, MBA, Study Chair — Paracelsus Medical University
Locations (1):
- Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University, Salzburg, Austria

REFERENCES:
- [Background] Flynn KE, Pina IL, Whellan DJ, Lin L, Blumenthal JA, Ellis SJ, Fine LJ, Howlett JG, Keteyian SJ, Kitzman DW, Kraus WE, Miller NH, Schulman KA, Spertus JA, O'Connor CM, Weinfurt KP; HF-ACTION Investigators. Effects of exercise training on health status in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1451-9. doi: 10.1001/jama.2009.457. PMID 19351942
- [Background] Niebauer J, Hambrecht R, Velich T, Hauer K, Marburger C, Kalberer B, Weiss C, von Hodenberg E, Schlierf G, Schuler G, Zimmermann R, Kubler W. Attenuated progression of coronary artery disease after 6 years of multifactorial risk intervention: role of physical exercise. Circulation. 1997 Oct 21;96(8):2534-41. doi: 10.1161/01.cir.96.8.2534. PMID 9355890
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- See also: Paracelsus Medical University Salzburg, Austria — http://www.pmu.ac.at/
- See also: Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University Salzburg, Austria — http://www.salk.at/sportmedizin.html